CLINICAL TRIAL: NCT05511337
Title: Effect of Control in Oxalate and Citrate Intake on Gut Microbiota Composition in Patients With Urolithiasis: Double-blind Randomized Clinical Study
Brief Title: Gut Microbiota in Patients With Urolithiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Regional de Alta Especialidad de la Península de Yucatán (Other)
Responsible Party: Principal Investigator, Azalia Avila Nava, PhD, Principal Investigator, Hospital Regional de Alta Especialidad de la Península de Yucatán
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2020-022
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Participants are randomized into three groups for 28 days:
  Control: caloric restriction or intervention A: Control oxalate and citrate foods or intervention B: Real-life intervention, control of oxalates and citrates without restriction of kilocalories.
  Randomization was performed by balanced blocks of three cells, with the research randomizer randomization program, 60 sites were randomized, which 20 participants were divided into three groups. Randomization was carried out by a person outside the study. Treatment will be given only through dietary counseling. Treatment adherence will be assessed in all groups through three food diaries (two on weekdays and one on weekends). Adherence will be considered if the participant complies with 80% of the treatment.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The person performing the measurements will be blinded to the group to which each participant belongs.
  The statistical analysis will be performed by a person who is blinded to the group to which the participants belong.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): Caloric restriction
  Interventions: Other: Caloric restriction
- Intervention A (Experimental): Caloric restriction and control oxalate and citrate food
  Interventions: Other: Caloric restriction and control oxalate and citrate foods
- Intervention B (Experimental): Real-life intervention, control of oxalates and citrates without restriction of kilocalories.
  Interventions: Other: Real-life intervention with control oxalate and citrate foods

INTERVENTIONS:
Other: Caloric restriction and control oxalate and citrate foods — Restriction of 500 kilocalories from the usual diet plus a decrease in oxalate-rich foods (< 40 mg per day) and an increase in citrate-rich foods (> 40 mEq per day) for 28 days. The treatment will be given through an individualized meal plan.
  Arms: Intervention A
Other: Caloric restriction — Restriction of 500 kilocalories from the usual diet for 28 days. The treatment will be given through an individualized meal plan
  Arms: Control
Other: Real-life intervention with control oxalate and citrate foods — Decrease in oxalate-rich foods (< 40 mg per day) and an increase in citrate-rich foods (> 40 mEq per day) without restriction in kilocalories from the usual diet for 28 days. Treatment will be given only through dietary counseling.
  Arms: Intervention B

SUMMARY:
Urolithiasis (UL) is the presence of kidney stones in different compartments such as ureters, bladder and/or urethra. Based on its incidence and prevalence it is considered a public health problem worldwide. In Mexico, especially in Yucatan state, is considered an endemic area of UL with a prevalence of 5.5%. There are several risk factors associated with the development of UL, among which are genetics, age, sex, excess weight, diet, and gut microbiota. In the diet there is promoters and inhibitors of stone formation, such as oxalates and citrates respectively. The gut microbiota is the set of microorganisms that inhabit the gastrointestinal tract, which have been related to the regulation of metabolic processes such as production of short-chain fatty acids (SCFA), vitamin K synthesis, and stimulation of the immune response. However, alterations in the composition of the microbiota have been associated with the development of various pathologies including UL. Recent studies have shown that the intestinal microbiota of people with kidney stones have a lower diversity and a different bacterial composition compared with healthy people, suggesting that interactions in the gut-renal axis could have a direct effect on the development of UL. Furthermore, these modifications could modulate oxalate and citrate transporters. Dietary modifications may decrease the risk of UL formation through increased consumption of citrate-rich foods (>40 mEq per day) and decreased consumption of oxalate-rich foods (< 40mg per day). It is known that dietary modifications can modulate the gut microbiota, however there is no evidence about the effect of a dietary intervention with oxalate and citrate control on the modulation of the microbiota in patients with UL. Thus, it is important to search for strategies to reduce UL, as well as the complications associated with them like chronic kidney disease. The main of the study is evaluate the effect of a dietary intervention with oxalate and citrate control on the composition and diversity of the intestinal microbiota of adults with UL.

DETAILED DESCRIPTION:
The protocol will be carried out in the Hospital Regional de Alta Especialidad de la Península de Yucatán (HRAEPY). This is double-blind randomized clinical study will be carried out in adults with a diagnosis of UL. Participants with UL are randomized by into three groups for 28 days. Control group: Caloric restriction, restriction of 500 kilocalories from the usual diet, or Intervention A: Restriction of 500 kilocalories from the usual diet plus a decrease in oxalate-rich foods (< 40 mg per day) and an increase in citrate-rich foods (> 40 mEq per day), or Intervention B: Real-life intervention with control oxalate and citrate foods: decrease in oxalate-rich foods (< 40 mg per day) and an increase in citrate-rich foods (> 40 mEq per day) without restriction of kilocalories from the usual diet. Randomization was performed by balanced blocks of three cells, with the research randomizer randomization program, 60 sites were randomized, which 20 participants were divided into three groups. Randomization was carried out by a person outside the study.

At the beginning and at the end of the interventions, the following characteristics will be determined anthropometric measurements (weight, height, waist circumference, body mass index (BMI)) and blood pressure. A 24-h urine sample is requested to determine oxalates and citrates. A fasting blood sample of 8-10 hours will be requested for the determination of the concentration of creatinine, uric acid, calcium, phosphorus and sodium. A stool sample will also be requested for DNA extraction, which will be used for analysis of the composition and biodiversity of the intestinal microbiota. The person performing of measurements will be blinded to the group to which each participant belongs. Treatment will be given only through dietary counseling. Follow-up is done by telephone monitoring once a week through logbook and reminders. At the end of the study, the statistical analysis will be performed by a person who is blinded to the group to which the participants belong.

The sample size was calculated with the formula for comparison of two proportions, with a one-tailed significance of 0.05 and a power of 80%, with a change in alpha diversity in the intervention group of 57% and in the control group of 18%. The result was 16 patients per group, but a 20% loss was considered. Therefore, a total of 20 participants per group was considered.

ELIGIBILITY:
Inclusion criteria:

* Subjects living in Merida, Yucatan
* Female or male
* Age between 18 and 60 years
* Confirmed diagnosis of UL confirmed with ultrasound (≥5mm) and/or radiographs or who had expelled a stone in a time no longer than 7 days at the time of selection
* BMI ≥ 25 and ≤ 39.9 kg/m2; no antibiotic intake (last 30 days)
* No intake of probiotics, prebiotics or synbiotics (last 15 days)
* No intake vitamin C supplements (last 15 days)
* No intake calcium supplements (last 15 days)

Exclusion criteria:

* Previous medical diagnosis of chronic kidney disease
* Serum creatinine >1.2 mg/dL
* Glomerular filtration <60 mL/min or 130 mL/min
* Type 2 diabetes
* Renal tubular acidosis
* Pregnancy

Elimination criteria:

* Not meeting 80% adherence to treatment
* Antibiotic consumption during the intervention

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Relative abundance of gut microbiota | At the beginning of the study and after 28 days of intervention
  Changes in relative abundance of phylum, gender and species of bacteria in gut microbiota

SECONDARY OUTCOMES:
Concentration of urinary citrate excretion | At the beginning of the study and after 28 days of intervention
  Changes in concentration of citrate excretion in 24-hour urine
Concentration of urinary oxalate excretion | At the beginning of the study and after 28 days of intervention
  Changes in concentration of oxalate excretion in 24-hour urine
Concentration of serum creatinine | At the beginning of the study and after 28 days of intervention
  Changes in concentration of creatinine in serum
Concentration of serum calcium | At the beginning of the study and after 28 days of intervention
  Changes in concentration of calcium in serum
Concentration of serum uric acid | At the beginning of the study and after 28 days of intervention
  Changes in concentration of uric acid in serum
Concentration of serum phosphorus | At the beginning of the study and after 28 days of intervention
  Changes in concentration of phosphorus in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Azalia Avila Nava, PhD, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Areses Trapote R, Urbieta Garagorri MA, Ubetagoyena Arrieta M, Mingo Monge T, Arruebarrena Lizarraga D. [Evaluation of renal stone disease: metabolic study]. An Pediatr (Barc). 2004 Nov;61(5):418-27. doi: 10.1016/s1695-4033(04)78417-9. Spanish. PMID 15530322
- [Background] Medina-Escobedo M, Zaidi M, Real-de Leon E, Orozco-Rivadeneyra S. [Urolithiasis prevalence and risk factors in Yucatan, Mexico]. Salud Publica Mex. 2002 Nov-Dec;44(6):541-5. Spanish. PMID 20383456
- [Background] Zuckerman JM, Assimos DG. Hypocitraturia: pathophysiology and medical management. Rev Urol. 2009 Summer;11(3):134-44. PMID 19918339
- [Background] Ticinesi A, Milani C, Guerra A, Allegri F, Lauretani F, Nouvenne A, Mancabelli L, Lugli GA, Turroni F, Duranti S, Mangifesta M, Viappiani A, Ferrario C, Dodi R, Dall'Asta M, Del Rio D, Ventura M, Meschi T. Understanding the gut-kidney axis in nephrolithiasis: an analysis of the gut microbiota composition and functionality of stone formers. Gut. 2018 Dec;67(12):2097-2106. doi: 10.1136/gutjnl-2017-315734. Epub 2018 Apr 28. PMID 29705728
- [Background] Del Chierico F, Vernocchi P, Dallapiccola B, Putignani L. Mediterranean diet and health: food effects on gut microbiota and disease control. Int J Mol Sci. 2014 Jul 1;15(7):11678-99. doi: 10.3390/ijms150711678. PMID 24987952
- [Background] Stanislawski MA, Frank DN, Borengasser SJ, Ostendorf DM, Ir D, Jambal P, Bing K, Wayland L, Siebert JC, Bessesen DH, MacLean PS, Melanson EL, Catenacci VA. The Gut Microbiota during a Behavioral Weight Loss Intervention. Nutrients. 2021 Sep 18;13(9):3248. doi: 10.3390/nu13093248. PMID 34579125
- See also: Manejo nutriológico en el paciente con litiasis renal — https://www.imbiomed.com.mx/articulo.php?id=110852